CLINICAL TRIAL: NCT05427617
Title: Clinical Application of Circulating Tumor DNA (ctDNA) to Guided the Late-Line Treatment for Patients With Late-Stage Breast Cancer
Brief Title: Circulating Tumor DNA (ctDNA)-Guided Late-Line Treatment in Patients With Late-Stage Breast Cancer
Acronym: ACTDNAGLT
Status: Completed | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYJJ-2020-022
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Breast Cancer; Circulating Tumor DNA; Gene Abnormality
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups; Diagnosis-Related Groups; Fulvestrant; Histone Deacetylase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood lymphocytes (PBL) and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Control group includes patients without ctDNA abnormality and patients without druggable ctDNA abnormality.
  Interventions: Drug: Control group
- Case group: Case group includes patients with druggable ctDNA abnormality.
  Interventions: Drug: Case group

INTERVENTIONS:
Drug: Control group — Physician chosen treatment
  Groups: Control group
Drug: Case group — Druggable ctDNA alterations-guided therapy
  Other Names: PARP inhibtior; EGFR inhibitor; CDK4/6 inhibitor; AR antagonists; anti-VEGFR; anti-FGFR; Fulvestrant; ADC drugs; PI3K inhibitor; anti-HER2 treatment; HDAC inhibitor
  Groups: Case group

SUMMARY:
This is a retrospective, observational, multi-center clinical study of circulating tumor DNA (ctDNA) to guide late-line therapy in late-stage metastatic breast cancer patients.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of plasma ctDNA mutation in guiding late-line treatment for late-stage metastatic breast cancer patients. Meanwhile, this study tries to evaluate the curative effect of ctDNA subtype-guided late-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Recent progression of TNBC after multiple lines of chemotherapy or of HR+ or HER2+ MBC after multiple lines of endocrine or targeted therapy;
* No available recommendation for the next treatment regimen;
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
* An updated, available pathological HR/HER2 status for metastasis;
* According to RECIST 1.1 standard, there should be at least one measurable target lesion;
* The expected survival time is > 3 months;
* Those aged 18-70 years old;
* Liver and kidney function and blood routine test meet the following conditions: Neutrophil > 2.0g/l, Hb > 9g / L, PLT > 100g / L; ALT and AST < 2.5ULN; TBIL < 1.5ULN; Cr < 1.0ULN
* Signing informed consent;
* Those willing to accept polygenic testing.

Exclusion Criteria:

* Patients with multiple primary tumors;
* Those who are unable to obtain blood samples;
* Those with a history of immunodeficiency or organ transplantation;
* Those with abnormal cardiac function or previous history of myocardial infarction or serious arrhythmia;
* The researchers think it is not suitable to participate in this experiment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study recruited consecutive patients with recent progression of metastatic TNBC after multiple lines of chemotherapy or of HR+ or HER2+ metastatic breast cancer after multiple lines of endocrine or targeted therapy.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | From the beginning of the treatment to the end of Cycle 2 (each cycle is 28 days) of treatment.
  The total rate of CR+PR+SD after the completion of two cycles of late-line therapy.
Progression-Free Survival | From date of recruitment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  The survival time between the beginning of treatment to death or the progression.

IPD SHARING:
Plan to Share IPD: No